CLINICAL TRIAL: NCT02423460
Title: Threonine Requirement in Healthy Adult Subjects and in Patients With Crohn's Disease and With Ulcerative Colitis Using the Indicator Amino Acid Oxidation (IAAO) Methodology
Brief Title: Threonine Requirement in IBD Adults and Healthy Adult Controls
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Collaborators: The Hospital for Sick Children (Other); Mount Sinai Hospital, Canada (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 1000046356
Record Dates: First submitted 2015-04-12; First posted 2015-04-22 (Estimated); Last update posted 2018-11-06 (Actual); Status verified 2018-11

CONDITIONS: Ulcerative Colitis; Crohn's Disease; Healthy
Keywords: Ulcerative Colitis; Healthy Controls; Crohn's Disease
MeSH Terms: conditions — Colitis, Ulcerative; Crohn Disease | interventions — Threonine; Amino Acids

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Threonine requirement (Experimental): The threonine requirement in healthy male subjects and in patients with Crohn's disease and Ulcerative colitis
  Interventions: Other: Threonine

INTERVENTIONS:
Other: Threonine — Threonine will be fed at various intake levels ranging from high to low in order to determine its requirement in healthy males and in patients with Crohn's disease and Ulcerative colitis.
  Other Names: amino acid

SUMMARY:
The daily requirement of threonine, an essential amino acid, will be evaluated in healthy adult males and in adult males with Crohn's Disease or ulcerative colitis using the indicator amino acid oxidation (IAAO) method. Participants will consume specially formulated diets with varying levels of threonine.

DETAILED DESCRIPTION:
Threonine is an essential amino acid which must be obtained from the diet. It is a component of mucin. Mucin, in turn, is a key protein in the mucous membrane that protects the lining of the intestine.

Inflammatory bowel disease (IBD) is a group of inflammatory conditions that affect the colon and small intestine. IBD primarily includes ulcerative colitis (UC) and Crohn's disease (CD). In UC, the inflammation is usually in the colon whereas in CD inflammation may occur anywhere along the digestive tract. Studies in animals have shown that more threonine is used when there is inflammation in the intestine.

The threonine requirement in healthy participants and in IBD patients will be determined using the indicator amino acid oxidation method. The requirement derived in healthy participants will be compared to that derived in patients with IBD.

Each participant will take part in two x 3 day study periods. The first two days are called adaptation days where the subjects will consume a liquid diet specially designed for him. The diet will be consumed at home. It contains all vitamins, minerals, protein and all other nutrients required. On the third day, the participant will come to the Hospital for Sick Children in Toronto. Subjects will consume hourly meals for a total of 8 meals and a stable isotope 13C-phenylalanine. Breath and urine samples will be collected to measure the oxidation of phenylalanine from which the threonine requirement will be determined.

ELIGIBILITY:
Inclusion Criteria (healthy controls):

* Male age 18 - 40 years of age
* Having obtained his (or his legal representative's) written informed consent.
* Normally nourished and without any inter-current illness.
* Absence of an active inflammatory process in the past month.

Exclusion Criteria (healthy controls):

* Subject who cannot be expected to comply with the study procedures.
* Currently participating or having participated in another clinical study during the last 4 weeks prior to the beginning of this study.

Inclusion Criteria: Crohn's Disease and Ulcerative Colitis

* Male age 18 - 40 years of age
* Having obtained his (or his legal representative's) Written Informed Consent.
* For both conditions, stable disease state and not malnourished per the treating physician.
* CD: Harvey Bradshaw Index (HBI) ≤ 8, disease location: evidence of ileal and or colon inflammatory involvement, no known strictures
* UC: Mayo Score ≤ 7 (or Partial Mayo Score ≤5)
* No tube feeding - Subjects must be treated and followed by the Gastroenterology team at Mt. Sinai Hospital, Toronto.

Exclusion Criteria: Crohn's Disease and Ulcerative Colitis

* Uncontrolled inflammation which will likely require surgery or escalation of therapy in the next 4 weeks
* Concomitant treatment:corticosteroids > 20mg/day
* Subject who cannot be expected to comply with the study procedures. - Subjects not treated and followed by the Gastroenterology team at Mt. Sinai Hospital, Toronto

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 86 (Actual)
Dates: Start 2015-05; Primary Completion 2018-09-17 (Actual); Study Completion 2018-09-23 (Actual)

PRIMARY OUTCOMES:
Threonine requirement in those with Crohn's Disease, ulcerative colitis and in healthy controls determined using the indicator amino acid oxidation method | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada